CLINICAL TRIAL: NCT07290426
Title: A Prospective Clinical Study Evaluating Pulse Dye Laser on Clearance of Vascular Indications
Brief Title: Vbeam Pro Pulse Dye Laser for the Treatment of Vascular Conditions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBP25005
Record Dates: First submitted 2025-12-16; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rosacea; Vascular Diseases; Port-Wine Stain
MeSH Terms: conditions — Rosacea; Vascular Diseases; Port-Wine Stain

STUDY DESIGN:
Intervention Model Description: Treatment Group with Vbeam Pro Pulse Dye Laser
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vbeam Pro Treatment Group (Experimental): Treatment with Vbeam Pro Laser System, up to eight (8) study treatments
  Interventions: Device: Vbeam Pro Laser Treatment

INTERVENTIONS:
Device: Vbeam Pro Laser Treatment — Treatment with Vbeam Pro Laser System

SUMMARY:
This is a clinical study to evaluate the safety and performance of the Vbeam Pro Laser System for the treatment of vascular indications, including rosacea and port wine stain birthmarks.

DETAILED DESCRIPTION:
Study Design This is a non-randomized, open-label clinical study evaluating clinical treatments with the Vbeam Pro system for the treatment of vascular indications, including rosacea and port wine stain birthmarks. There are two phases of this study:

Phase I: Safety

1. Screening and Enrollment Visit
2. Up to Three (3) Treatment Visits (with treatment intervals from 2 weeks to 6 weeks).
3. 7 Day (+/- 5 days) Follow Up Visit following Each Treatment Session (may be a virtual telephone or video visit)
4. Additional follow-up visits may be required per the discretion of the principal investigator to assess safety and healing progression

Phase II: Safety, Efficacy, and Optimization of Treatment Parameters

1. Screening and Enrollment Visit
2. Treatment visits are limited to up to eight (8) study treatments (with treatment intervals from 1 week to 8 weeks).
3. Follow-up #1 (4 weeks - 8 weeks)
4. Follow-up #2 (8 weeks - 16 weeks) (optional)

Additional follow up visits may be added, if necessary, per Sponsor and investigators' discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 years or older
2. Presence of one or more vascular lesion, cutaneous lesion, or other dermatological condition deemed fit for treatment
3. Able and willing to comply with the treatment/follow-up schedule and comply with all study (protocol) requirements.
4. Willing to provide signed, informed consent to participate in the study
5. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications, presentations, and marketing materials

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months prior to enrollment into the study, and/or breast feeding
2. Known photosensitivity to 595nm or 1064 nm light
3. History of light-induced seizure disorders
4. Severe unstable concurrent conditions, such as unstable cardiac disorders
5. Use of implanted medical device including pacemakers, cardioverters and other implantable devices or fillers per investigator discretion (consultation with physicians prior to treatment is required)
6. Use of photosensitizing medications (medications that introduce photosensitivity or medications within or above the 595 nm wavelength, refer to Candela's list of drugs that may cause photosensitivity)
7. Tattoos (including decorative, permanent makeup and radiation port tattoos) in the intended study treatment area (595nm use only)
8. Active Herpes Simplex Virus (HSV) in the intended treatment area unless treated with prophylactic medication
9. The intended treatment area has significant sun exposure within the past 2 weeks or self-tanner has been applied to the treatment area
10. In the opinion of the Investigator, the subject is unwilling or unable to adhere to the study requirements or is otherwise unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clearance of Vascular Lesion | Baseline to Follow-up #1 (up to 72 weeks)
  Evaluation of clearance of vascular indications following treatment series as indicated by a minimum 1-point improvement on the validated Investigator's Global Assessment (IGA) Scale at study endpoint relative to baseline as rated by the principal investigator.

SECONDARY OUTCOMES:
Investigator Global Aesthetic Improvement Scale | Baseline to Follow-up #1 (up to 72 weeks)
  Evaluation of investigator rated scales following the treatment series Evaluation of investigator GAIS following the treatment series for treatment areas or comparing split treatment areas
Subject Satisfaction Scale | Baseline to Follow-up #1 (up to 72 weeks)
  Evaluation of subject satisfaction following the treatment series for treatment areas or comparing split treatment areas.

IPD SHARING:
Plan to Share IPD: No